CLINICAL TRIAL: NCT01199354
Title: Phase II Study: Assessing the Feasibility and Morbidity of Skin Sparing Mastectomy and Immediate Breast Reconstruction With Latissimus Dorsi Flap After Neoadjuvant Chemotherapy and Radiotherapy in Invasive Breast Carcinoma.
Brief Title: Skin Sparing Mastectomy and Immediate Breast Reconstruction With Latissimus Dorsi Flap After Neoadjuvant Chemotherapy and Radiotherapy (M-RIC)
Acronym: M-RIC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinique Clementville (Other)
Responsible Party: Jean-Louis Bonneton, Clinique Clementville
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CLEM-01
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Breast Carcinoma
Keywords: Invasive breast carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy

INTERVENTIONS:
Procedure: Mastectomy, preservation of the skin envelope,followed by immediate reconstruction with autologous latissimus dorsi flap. — Mastectomy, preservation of the skin envelope, removal of the nipple-areolar complex and dissection of the axillary lymph nodes followed by immediate reconstruction with autologous latissimus dorsi flap with or without prosthesis.

SUMMARY:
The aim of the study is to evaluate the feasibility and morbidity of skin sparing mastectomy and immediate breast reconstruction with latissimus dorsi flap after neoadjuvant chemotherapy and radiotherapy in invasive breast carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Women < 75 year old
* Invasive breast carcinoma, indication for mastectomy
* Women Health Organization (WHO) score of 0 and 1, primary chemotherapy, external radiotherapy performed less than 8 week earlier...

Exclusion Criteria:

* Women older than 75
* Metastatic breast carcinoma
* Antecedents of previously treated homolateral breast carcinoma
* Documented cancer progression
* Smoker at the moment of the indication surgery
* Known diabetes, neoadjuvant hormonal treatment...

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-07; Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of skin necrosis
  To evaluate the incidence of skin necrosis in case of treatment with skin sparing mastectomy and immediate breas reconstruction with latissimus dorsi myocutaneous flap after neoadjuvant chemotherapy and radiotherapy.

SECONDARY OUTCOMES:
Rate of histological remission of the surgical specimen based on the anatomopathological examination

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Zinzindhoue, Principal Investigator — Clinique Clementville
Locations (9):
- France (9):
  - Polyclinique Urbain V, Avignon
  - Centre Jean Perrin, Clermont-Ferrand
  - Groupe Hospitalier Mutualiste Clinique les Eaux Claires, Grenoble
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Clinique Clementville, Montpellier
  - CRLCC Val d'Aurelle, Montpellier
  - Clinique Belledonne, Saint-Martin-d'Hères
  - Institut Claudius Regaud, Toulouse